CLINICAL TRIAL: NCT07166783
Title: Pharmacokinetics, Pharmacological Effects and Safety of Single Dose of 7.5mg Tolvaptan Tablet in Healthy Male Subjects
Brief Title: Single Dose of 7.5mg Tolvaptan Phase I Clinical Trial Protocol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-11-807-01
Record Dates: First submitted 2025-08-22; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Health Subjects
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 7.5mg Tolvaptan single dose (Experimental)
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — single dose oral administration of 7.5mg Tolvaptan

SUMMARY:
Pharmacokinetics, pharmacological effects and safety of single dose of 7.5mg Tolvaptan tablet in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male, signing the informed consent form;
2. At the time of signing the informed consent form, aged between 18 and 40 years old (inclusive);
3. Body weight no less than 50kg, body mass index within the range of 19 to 24 (inclusive);
4. Proven to be a healthy subject based on the results of medical history, serological tests (HIV antibody, HBsAg, HCV antibody and syphilis antibody), physical examination, vital signs (temperature, blood pressure, pulse), 12-lead electrocardiogram, and laboratory tests (blood routine, blood biochemistry, coagulation function and urine routine).

Exclusion Criteria:

1. Those with a history of heart, liver, kidney, digestive tract, metabolic disorders, respiratory, blood, mental or nervous system diseases, or those judged by the physician as unsuitable.
2. Those with a history of clinically significant arrhythmias of any type, including a family history of genetic diseases (relatives with a history of arrhythmias with genetic predisposition), such as rapid and slow types, including atrioventricular block, sinus arrest, supraventricular tachycardia, etc.
3. Those with a history of drug or other substance allergies, allergic constitution or tendency.
4. Those known to be intolerant to the components of the test drug (including lactose), such as those with rare hereditary galactose intolerance, lactase deficiency or glucose-galactose malabsorption.
5. Those with various urinary disorders (such as frequent urination or difficulty in urination, etc.).
6. Those who smoke, are alcoholics or have other drug dependencies.
7. Those who have donated blood or lost an equivalent amount of blood (>350 ml) within 12 weeks before enrollment.
8. Those who have participated in any drug trials within 12 weeks before enrollment.
9. Those who have taken any preventive or therapeutic drugs within the past 2 weeks.
10. Those who have consumed grapefruit or grapefruit-containing foods within one week before taking the drug.
11. Those whose diet is significantly deviated from normal protein, carbohydrate and fat intake as judged by the investigator (such as vegetarians or absolute vegetarians).
12. Those with a history of orthostatic hypotension (a drop in blood pressure of ≥20/10 mmHg when changing from a lying to a standing position, accompanied by symptoms such as dizziness), orthostatic dizziness, syncope, fainting or vertigo.
13. Those whose resting pulse rate is less than 55 beats per minute or more than 90 beats per minute after sitting quietly for more than 3 minutes.
14. Those whose sitting systolic blood pressure is less than 100 mmHg or more than 140 mmHg, or whose diastolic blood pressure is less than 60 mmHg or more than 90 mmHg after sitting quietly for more than 3 minutes.
15. Those with clinically significant 12-lead electrocardiogram changes.
16. Those with clinically significant physical examination abnormalities.
17. Those with positive results for HIV antibody, HBsAg, HCV antibody or syphilis antibody tests.
18. Other conditions judged by the researcher as potentially affecting the subject's completion of the trial.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06-16 (Actual); Primary Completion 2011-07-04 (Actual); Study Completion 2011-07-04 (Actual)

PRIMARY OUTCOMES:
Tolvaptan PK parameter | On Day 1 pre-dose and post-dose 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours.
  peak concentration (Cmax)
Tolvaptan PK parameter | On Day 1 pre-dose and post-dose 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours
  time to peak (Tmax)
Tolvaptan PK parameter | On Day 1 pre-dose and post-dose 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours
  area under the drug-time curve (AUC0-t and AUC0-∞)
Tolvaptan PK parameter | On Day 1 pre-dose and post-dose 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours
  elimination half-life (t1/2)
Tolvaptan PK parameter | On Day 1 pre-dose and post-dose 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours
  apparent clearance (CL/F)
Tolvaptan PK parameter | On Day 1 pre-dose and post-dose 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours
  apparent volume of distribution (Vd/F)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Liu H, Liu T, Liu M, Zheng X, Zhong W, Zhao Q, Jiang J, Hu P, Li Y. Clinical trial on the pharmacokinetics, pharmacodynamics and safety of tolvaptan in healthy Chinese males: an open-label, single and multiple dosage, parallel group study. Front Pharmacol. 2025 Nov 21;16:1713702. doi: 10.3389/fphar.2025.1713702. eCollection 2025. PMID 41357896